

| nitials: | Date: |
|----------|-------|



Institutional Review Board
1204 Marie Mount Hall ● 7814 Regents Drive ● College Park, MD 20742 ● 301-405-4212 ● <u>irb@umd.edu</u>

## **CONSENT TO PARTICIPATE**

| Project Title | Effects of Youth Mental Health First Aid (YMHFA) on South Asian |
|---|---|
| | American Adults working with South Asian American Youth |
| Purpose of the Study | This research is being conducted by <b>Ami Patel, M.A</b> and <b>Dr. Cixin Wang, Ph.D.</b> at the University of Maryland, College Park. We are inviting you to participate in this research project because you are participating in YMHFA training. The purpose of this research project is to examine the efficacy of the YMHFA training with South Asian American adult participants (18 years or older) who are working with South Asian American youth. |
| Procedures | You will be invited to participate in an interview to provide suggestions about how to modify YMFHA to better serve South Asian American youth. Your suggestions will help us improve the YMHFA training. |
| | You will participate in <b>one of two</b> groups to receive the YMHFA training. If you take the first training, <u>you will be asked to complete a survey two times</u> . It will be the same survey each time, and it should take about 20 minutes to complete it each time. |
| | If you take the second training, <u>you will be asked to complete the survey three times</u> . It will be the same survey each time, and it should take about 20 minutes to complete it each time. |
| | The survey includes measures that assess stigma, knowledge of mental health, confidence in helping, intentions to implement the five-step action plan, implementation of the plan (at post-training), acceptability of the intervention, etc. All adults who attend YMHFA are invited to participate in this research. |
| | We invite participants to complete the <u>same</u> survey over time to help us evaluate the effectiveness of the training. |
| | Additionally, you <u>may</u> be invited to participate in a focus group after completion of the training and surveys to gather your feedback about the training to help us improve future trainings. |
| Potential Risks and Discomforts | There are no risks for completing the research component of the project. |
| | During the YMHFA training, there will be ample opportunities to take breaks and debrief after discussing serious topics related to mental health. A co-facilitator on the University of Maryland team is a licensed psychologist and will be available if participants would like to talk more after the training about any discomfort or concerns. Additionally, a list of mental health resources will be provided to all training participants as part of the training. |

IRBNet Package: 1366194-26 Page 1 of 3

| nitials: | Date: |
|----------|------------|
| muaio. | <br>Duito. |

| Potential Benefits | There are no direct benefits to the individuals for participating in this |
|---|---|
| l otential Benefits | research study. However, we expect participants who participate in |
| | the training to gain a better understanding of how to help adolescents |
| | who are experiencing mental health concerns or crises. We hope |
| | that, in the future, other people might benefit from this study through |
| | new understanding of how the YMHFA training can be improved. |
| Confidentiality | Any potential loss of confidentiality will be minimized by storing |
| | electronic data (e.g., demographic information and survey data, and |
| | the audio recording of any interviews, as applicable) on password |
| | protected computers. Any potential loss of confidentiality will also be |
| | minimized by assigning all participants an ID number and only using |
| | this number to identify you on survey measures. All data are entered |
| | and stored using a coded identification number: (1) Participants' |
| | name will not be included in the data file; (2) a code will be placed on |
| | the survey; (3) through the use of an identification number, the PI will |
| | be able to link the survey to participant's identity; and (4) only the PI |
| | will have access to the list of identification numbers. This list will be |
| | destroyed once all data have been collected. |
| | If we write a report or article about this research project, your identity |
| | will be protected to the maximum extent possible. Your information |
| | may be shared with representatives of the University of Maryland, |
| | College Park or governmental authorities if you or someone else is in |
| | danger or if we are required to do so by law. |
| Compensation | Participants who sign up to complete the full 5.25-hour training will |
| | receive access to the training manual and other course materials for |
| | free. |
| | You will receive up to a \$30 e-gift card via email for completing all |
| | surveys. |
| | Any suspected fraud or abuse will result in forfeiture of |
| | compensation. |
| Right to Withdraw | Your participation in this research is completely voluntary. You may |
| and Questions | choose not to take part at all. If you decide to participate in this |
| | research, you have the option to stop participating at any time. If you |
| | decide not to participate in this study or if you stop participating at any time, you will not be penalized or lose any benefits to which you |
| | otherwise qualify. |
| | otherwise quality. |
| | If you are an employee or student at the University of Maryland, your |
| | employment status or academic standing will not be positively or |
| | negatively affected by your participation or non-participation in this |
| | study. |
| | If you wish to stop taking part in the study, or if you have questions, |
| | concerns, complaints, and/or or if you need to report an injury related |
| | to the research, please contact the investigator: |
| | Ami Patel |
| | amikumar@umd.edu If you have questions about your rights as a research participant or |

| nitials: | Date: |
|----------|-------|

| | wish to report a research-related injury, please contact: |
|---|---|
| | University of Maryland College Park |
| | Institutional Review Board Office |
| | 1204 Marie Mount Hall |
| | College Park, Maryland, 20742 |
| | E-mail: irb@umd.edu |
| | Telephone: 301-405-0678 |
| | For more information regarding participant rights, please visit: |
| | https://research.umd.edu/irb-research-participants |
| | This research has been reviewed according to the University of Maryland, College Park IRB procedures for research involving human |
| | subjects. |
| Statement of Consent | |
| | You may request a copy of this consent form by emailing amikumar@umd.edu. |
| | If you agree to participate, please provide your name and date below. |
| Signature and Date (provided | NAME OF PARTICIPANT |
| electronically) | SIGNATURE OF PARTICIPANT |
| | DATE |